CLINICAL TRIAL: NCT00139880
Title: A Single Center, Randomized, Double-blind, Crossover Pilot Trial Comparing the Onset of Action of Parcopa™ With Sinemet® in Subjects With Stable Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SP867
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

INTERVENTIONS:
Drug: Parcopa

SUMMARY:
To test whether Parcopa, a new Orally Disintegrating Tablet of Carbidopa-Levodopa, has a faster onset of action, changes in the UPDRS Motor Exam score at intervals after a single dose of Parcopa or Sinemet are being compared in 10 subjects with Parkinson's disease. Subjects 40 years or older having idiopathic PD with Hoehn and Yahr state II or III are eligible if taking a stable dose of < 200 mg carbidopa and < 2000 mg levodopa daily. At both treatment visits, either Parcopa or Sinemet, plus a placebo of the opposite tablet (ODT or conventional) are administered. The dose is the same as the subject's prestudy regimen. The primary efficacy variable, time to onset of action, is the first postdose time when a 30% decrease (30% improvement) in the total score is achieved. All UPDRS evaluations are done by a rater blinded to the active treatment received by the subject.

DETAILED DESCRIPTION:
See approved Package Insert for Adverse Event information.

ELIGIBILITY:
Inclusion Criteria:

* Stable Parkinson's disease

Exclusion Criteria:

* idiopathic PD with Hoehn and Yahr state II or III

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States